CLINICAL TRIAL: NCT06797856
Title: Measurement of Refractive Error in Pseudophakic Eyes Using an Autorefractor and a Wavefront Aberrometer
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDEV112ARGS
Record Dates: First submitted 2025-01-27; First posted 2025-01-29 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Measurement of Refractive Error

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Refractive Error: * Refractive error centrally (on-axis) and peripherally in both nasal and temporal visual fields
  * Ocular wavefront measured centrally (on-axis) and peripherally in both nasal and temporal visual fields
  Interventions: Diagnostic Test: Refractive Error

INTERVENTIONS:
Diagnostic Test: Refractive Error — * Refractive error centrally (on-axis) and peripherally in both nasal and temporal visual fields
  * Ocular wavefront measured centrally (on-axis) and peripherally in both nasal and temporal visual fields

SUMMARY:
Prospective, single-site, non-interventional, technician masked, randomized (instrument and examiner testing sequences), controlled, bilateral, parallel-group study.

ELIGIBILITY:
Inclusion Criteria following Screening

The subject must:

1. Read, understand, and sign the Statement of Informed Consent and HIPAA authorization and receive a fully executed copy of the form(s).
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be 40 years of age or older at the time of enrollment.
4. Be pseudophakic in at least one eye, with that eye (hereafter referred to as the 'study eye') implanted with either the TECNIS Eyhance™ IOL (model ICB00, GIB00 or DIB00) or the TECNIS® Monofocal 1-Piece IOL (model ZCB00 or DCB00).
5. Have had IOL surgery for the study eye completed at least 3 months prior to enrollment, with enough time elapsed between surgery and enrollment such that the refraction has stabilized in that eye.

   Inclusion Criteria at Baseline Evaluation

   The subject must:
6. In the study eye, meet the following criteria with regard to the non-vertex-corrected (i.e., spectacleplane) distance subjective refraction:

   1. Mean spherical equivalent must be between +2.00 and -2.00 DS (inclusive).
   2. The magnitude of the cylinder must be 1.50 DC or less.
7. Have best-corrected visual acuity of at least 20/32 in the study eye.

Exclusion Criteria following Screening

The subject must not:

1. Be pregnant.
2. Have uncontrolled diabetes by self-report.
3. Have a history of ocular trauma, systemic disease or medication use known to cause variability in refractive error.
4. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.) other than bilateral cataract surgery with IOL implantation and YAG laser capsulotomy.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, scleral lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 3 months.
6. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site or study Sponsor.
7. Be taking any ocular or systemic medications known to adversely affect vision or cause miosis, or that may otherwise compromise study endpoints.
8. Be currently participating in or have participated in any other clinical trial within 30 days prior to enrollment. Exclusion Criteria at Baseline Evaluation

   The subject must not:
9. Have clinically significant slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities, or bulbar injection) or other corneal or ocular disease or abnormalities that, in the opinion of the investigator, may compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, corneal scar or opacity ≥ 0.3 mm, recurrent corneal erosions, moderate or above corneal distortion, herpetic keratitis).
10. Have posterior capsular opacification (PCO) that, in the opinion of the investigator, is significant enough that it is likely to detrimentally affect autorefraction or wavefront measurements. 11. Have fluctuations in vision due to clinically significant dry eye. 12. Have a history of strabismus, amblyopia, nystagmus, or any condition that affects fixation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 40 years of age or older who have been bilaterally implanted with either the TECNIS® Eyhance™ IOL (model ICB00, GIB00 or DIB00) or the TECNIS® Monofocal 1-Piece IOL (model ZCB00 or DCB00).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Refractive Error | Two study visits, 1 to 14 calendar days apart. Study duration approximately 6 months.
  * Refractive error centrally (on-axis) and peripherally in both nasal and temporal visual fields
  * Ocular wavefront measured centrally (on-axis) and peripherally in both nasal and temporal visual fields

CONTACTS AND LOCATIONS:
Locations (1):
- SoCal Eye, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu